CLINICAL TRIAL: NCT01548456
Title: Intramedullary Nailing Versus Plates for Femoral Shaft Fractures in Dar es Salaam, Tanzania With Minimum 1-Year Follow-up
Brief Title: Nails Versus Plates for Femur Fractures in Dar es Salaam, Tanzania
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Orthopaedic Research Foundation (Other); Orthopaedic Trauma Association (Other); Muhimbili Orthopaedic Institute (Other)
Responsible Party: Sponsor
Other Study IDs: UCSF 23346
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Femoral Fractures
Keywords: femur fracture; internal fixation; intramedullary nailing
MeSH Terms: conditions — Femoral Fractures | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intramedullary nailing: Subjects with a femur fracture who undergo operative fixation with an intramedullary nail
  Interventions: Procedure: Intramedullary Nailing
- Open Reduction Internal Fixation: Subjects with a femur fracture who undergo open reduction internal fixation with a dynamic compression plate
  Interventions: Procedure: Open Reduction Internal Fixation

INTERVENTIONS:
Procedure: Intramedullary Nailing — Surgical treatment that includes closed or open reduction and stabilization of the femur fracture with an intramedullary rod inserted using antegrade or retrograde technique
  Other Names: SIGN Intramedullary Nail
  Groups: Intramedullary nailing
Procedure: Open Reduction Internal Fixation — Surgical treatment that includes open reduction internal fixation of the femur fracture with a dynamic compression plate
  Groups: Open Reduction Internal Fixation

SUMMARY:
This is a prospective observational study of patients with femur fractures in Dar es Salaam, Tanzania comparing two different surgical techniques: intramedullary nailing (IMN) and open reduction internal fixation (ORIF) with a plate. The primary outcome is the rate of reoperation for any reason, and the secondary outcomes are fracture healing, return to work, and health-related quality-of-life. The investigators hypothesize that there will be a difference in the rate of reoperation for patients with femur fractures treated with an IMN compared to ORIF with a plate.

DETAILED DESCRIPTION:
The study will be a prospective clinical trial conducted at Muhimbili Orthopaedic Institute (MOI) in Dar es Salaam, Tanzania. All adult patients with diaphyseal femur fractures meeting the eligibility criteria will be invited to enroll. Study subjects will be treated at the discretion of the surgeons at MOI. This could include an intramedullary nail, a plate, external fixation, or skeletal traction. Potential confounders recorded will be age, gender, body mass index, comorbidities, fracture pattern, open versus closed injury, time from injury to presentation, time from presentation to surgery, and associated injuries. The primary outcome considered will be reoperation for any reason. Secondary outcomes will be clinical union, defined as full-painless weight bearing on the injured extremity, radiographic union, return to work, and health-related quality-of-life. Follow up will be scheduled at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year after surgery and will include both clinical and radiographic evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Diaphyseal fracture amenable to operative fixation with an intramedullary nail or plate
2. Age 18 to 65

Exclusion Criteria:

1. Clinical evidence of infection at the surgical site (defined clinically as drainage or erythema)
2. Pathologic fracture
3. Prior surgery
4. Presentation 3 weeks or more after injury
5. Inability or unwillingness to comply with follow up to 1-year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with diaphyseal fractures of the femur presenting to Muhimbili Orthopaedic Institute in Dar es Salaam, Tanzania will be considered eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Reoperation | 1-year
  Reoperation involving the affected femur for any reason within the first year will be considered an event.

SECONDARY OUTCOMES:
Health-related quality of life | 1-year
  Health-related quality of life as measured by the EQ-5D-3L (Swahili version) by the Euroqol Group
Return to work | 1-year
  Time from surgery to return to work among patients employed at the time of injury
Clinical union | 1-year
  Defined as full painless weight bearing on the affected extremity
Radiographic Union | 1-year
  Bony healing as measured by the Radiographic Union Scale in Tibial Fractures (RUST) Score

CONTACTS AND LOCATIONS:
Overall Officials: David W Shearer, MD, MPH, Principal Investigator — University of California, San Francisco; Edmund N Eliezer, MD, Study Director — Muhimbili Orthopaedic Institute
Locations (1):
- Muhimbili Orthopaedic Institute, Dar es Salaam, Tanzania